CLINICAL TRIAL: NCT07193680
Title: Angiogenic Markers for Confirming Term Preeclampsia (noPE-37 Trial): An Open-Label, Randomized Controlled Trial
Brief Title: NOPE37: Angiogenic Factors for Managing Term Preeclampsia
Acronym: NOPE37
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR(AMI)392-2023
Record Dates: First submitted 2025-07-21; First posted 2025-09-26 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Preeclampsia
Keywords: preeclampsia; angiogenic factors; expectant management
MeSH Terms: conditions — Pre-Eclampsia | interventions — Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care: elective delivery at 37 weeks of gestation (Active Comparator): In the control group, a blood test to assess the sFlt-1/PlGF ratio will be performed, and the result will be concealed from investigators. As in current clinical practice, elective delivery will be scheduled at 37 weeks. If preeclampsia is first diagnosed after 37 weeks, immediate delivery will be recommended. If at any time after enrollment any of the following is present, immediate delivery (within 24 hours) will be recommended: preeclampsia with severe features according to ACOG criteria, decreased fetal movements, absent or reversed diastolic flow in the umbilical artery, non-reassuring CTG, biophysical profile score ≤6, or oligohydramnios.
  Interventions: Other: Standard care: elective delivery at 37 weeks of gestation
- Intervention arm: expectant management if sFlt-1/PlGF<38 (Experimental): If sFlt-1/PlGF <38, expectant management will be followed until 39 weeks. If any other medical condition is present, local protocols for the specific condition will be followed. If fetal growth restriction in present (with antegrade diastolic umbilical flow), weekly repetition of sFlt-1/PlGF wil be done. If sFlt-1/PlGF ≥38, delivery at 37 weeks will be recommended, or immediate delivery if the patient is enrolled after 37 weeks. If at any time after enrollment any of the following is present, immediate delivery (within 24 hours) will be recommended: preeclampsia with severe features according to ACOG criteria, decreased fetal movements, absent or reversed diastolic flow in the umbilical artery, non-reassuring CTG, biophysical profile score ≤6, sFlt-1/PlGF ≥38 or oligohydramnios.
  Interventions: Other: Intervention arm: expectant management if sFlt-1/PlGF<38

INTERVENTIONS:
Other: Intervention arm: expectant management if sFlt-1/PlGF<38 — If the angiogenic factors are normal (sFlt-1/PlGF <38), expectant management will be followed until 39 weeks, instead of delivery at ≥37 weeks of gestation as in standard care for preeclampsia without severe features.
  Arms: Intervention arm: expectant management if sFlt-1/PlGF<38
Other: Standard care: elective delivery at 37 weeks of gestation — In the control arm, standard care for preeclampsia without severe features will be followed: elective delivery at ≥37 weeks of gestation.
  Arms: Standard care: elective delivery at 37 weeks of gestation

SUMMARY:
This study tests the hypothesis that, in women with preeclampsia without severe features, delivery management based on sFlt-1/PlGF would reduce the rate of induction of labor without worsening the rate of progression to preeclampsia with severe features and other maternal complications.

DETAILED DESCRIPTION:
Participants with preeclampsia without severe features between 36 and 38+6 weeks, who do not meet any exclusion criteria, will be randomly assigned to two groups:

* In the study group, if angiogenic factors are normal (sFlt-1/PlGF <38), delivery will be delayed until 39 weeks; if any other medical condition is present, delivery will be scheduled according to the specific protocol for it.
* In the study group, if angiogenic factors are abnormal (sFlt-1/PlGF ≥38), labor will be induced at ≥37 weeks.
* In the control group, labor will be recommended at 37 weeks, as is currently standard.
* In both groups, NT-proBNP levels will be measured at enrollment.
* In both groups, a satisfaction questionnaire will be completed at enrollment and 4 weeks after delivery.
* In both groups, if any of the following is present, delivery will be recommended immediately (within 24 hours):

  1. preeclampsia with severe features according to ACOG criteria
  2. decreased fetal movements
  3. absent or reversed diastolic flow in the umbilical artery
  4. non-reassuring CTG
  5. biophysical profile score ≤6
  6. oligohydramnios (largest vertical pocket <2 cm)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Singleton pregnancy
* Preeclampsia without severe features according to the ACOG definition
* Antegrade diastolic flow in the umbilical artery Doppler
* Gestational age between 36+0 and 38+6 weeks of gestation
* Gestational age confirmed by fetal crown-rump length measurement in the first-trimester scan (from 11+0 to 13+6 weeks of gestation) or by in vitro fertilization dates

Exclusion Criteria:

* Fetal death
* Preeclampsia with severe features according to the ACOG definition, eclampsia, or any condition that requires immediate delivery
* Absent or reversed end-diastolic flow in the umbilical artery Doppler
* Non-reassuring CTG
* Decreased fetal movements
* Biophysical profile score ≤6
* Oligohydramnios
* Refusal to provide informed consent
* Fetal malformation
* Placental abruption
* Antiphospholipid antibody syndrome

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2025-12-04 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Composite maternal outcome | through study completion, an average of 2 months
  The primary outcome is a composite poor maternal outcome, defined as maternal mortality, severe maternal morbidity (eclampsia, HELLP syndrome, thromboembolic disease, pulmonary edema, or placental abruption), preeclampsia with severe features, and major postpartum hemorrhage (>1000 mL).

SECONDARY OUTCOMES:
Neonatal morbidity | through study completion, an average of 2 months
  Neonatal morbidity is defined as the occurrence of at least one of the following: 5-minute Apgar score <7, NICU admission, fetal death, neonatal death, sepsis, hypoglycemia, transient tachypnea of the newborn, respiratory distress syndrome, meconium aspiration syndrome, periventricular leukomalacia, intraventricular hemorrhage, seizures, necrotizing enterocolitis, neonatal jaundice requiring phototherapy, neonatal birthweight <2500 g, or elective early-term delivery (37+0-38+6 weeks of gestation).
Method of delivery | through study completion, an average of 2 months
  Method of delivery, onset of labor, operative vaginal delivery for fetal distress, cesarean section for fetal distress.
Maternal admission to ICU | through study completion, an average of 2 months
  Maternal admission to ICU (yes/no)
Days of maternal admission to ICU | through study completion, an average of 2 months
  Duration of maternal admission to ICU (days)
Gestational age at delivery | through study completion, an average of 2 months
  Gestational age at delivery (weeks and days)
Birthweight | through study completion, an average of 2 months
  Birthweight in grams
Birthweight percentile | through study completion, an average of 2 months
  Birthweight percentile (%) according to local reference charts
Prematurity | through study completion, an average of 2 months
  Prematurity (delivery <37 weeks of gestation), yes/no
Days of neonatal admission to NICU | through study completion, an average of 2 months
  duration of neonatal admission to NICU (days)
Metabolic acidosis | through study completion, an average of 2 months
  Umbilical artery pH <7.10 and base excess <-12 mmol/L (yes/no)
Need of maternal corticosteroids | through study completion, an average of 2 months
  Need of maternal corticosteroids (yes/no)
Maternal NT-proBNP levels | through study completion, an average of 2 months
  Maternal NT-proBNP levels (pg/mL)
Maternal satisfaction measured by the Generic Short Patient Experiences Questionnaire (GS-PEQ) | through study completion, an average of 2 months
  Ten-item measure scored 1-5 per item (total range 10-50; higher scores = better patient experiences).

CONTACTS AND LOCATIONS:
Locations (23):
- Spain (23):
  - Hospital Universitari Dexeus, Barcelona, BARCELONA
  - Hospital Universitario de A Coruña, A Coruña
  - Hospital General Universitari Dr. Balmis, Alicante
  - Vall d'Hebron Hospital Campus, Barcelona
  - Hospital Universitario de Cabueñes, Cabueñes
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital General Universitario de Elche, Elche
  - Hospital Universitario de Getafe, Getafe
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona
  - Hospital Universitario San Cecilio, Granada
  - Hospital Universitario de Jerez, Jerez de la Frontera
  - Hospital Materno Infantil de Gran Canaria, Las Palmas de Gran Canaria
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital universitario 12 de Octubre, Madrid
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitari Son Espases, Palma de Mallorca
  - Hospital Universitario Virgen de Valme, Seville
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitari de Tarragona Joan XXIII, Tarragona
  - Consorci Sanitari de Terrassa, Terrassa
  - Hospital Universitari MútuaTerrassa, Terrassa
  - Hospital Universitario de Torrejón, Torrejón
  - Hospital Universitario Lozano Blesa, Zaragoza